CLINICAL TRIAL: NCT06969456
Title: Patient-centered Management of Chronic Spinal Pain by Addressing the Peripheral and Central Component With Exercise and Non-invasive Neuromodulation: A Randomized Control Trial (RCT)
Brief Title: Managing Chronic Spinal Pain With Exercise and Neuromodulation
Acronym: UCV/PSPS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Universidad Católica de Valencia San Vicente Mártir (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UCV/2024-2025/031
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-04

CONDITIONS: Spinal Pain Syndrome; Chronic Pain (Back / Neck)
Keywords: Chronic spinal pain; neuromodulation; motor control exercises; biopsychosocial approach; disability; quality of life
MeSH Terms: conditions — Chronic Pain | interventions — Exercise; Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The guidelines and treatment protocols will be overseen by the principal investigator and a team of specialist physiotherapists, each with over 10 years of experience in the management of neuromodulation and exercise therapy for chronic lumbar pain. Stratified randomization will be implemented to ensure that the compared groups are balanced with respect to the level of neuropathic pain. Prior to the randomization process, the baseline level of neuropathic pain shall be identified. Two strata of participants will be established within their own group. Subgroup 1 will include those participants who are on the DN4 scale of a value of 4,5,6 or 7. In subgroup 2 will be patients who are on the DN4 scale of a value of 8,9 or 10.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise + TDCS (Experimental): The transcranial direct current stimulation (tDCS) group will undergo 20 minutes of continuous stimulation at an intensity of 1.5 mA over the left dorsolateral prefrontal cortex (DLPFC) during each session. Two saline-soaked sponge electrodes, each measuring 35 cm², will be utilized. In accordance with the international 10-20 EEG electrode placement system, the anodal electrode will be positioned over F3 to specifically target the left DLPFC. The reference electrode will be placed over the left eye to ensure that the current traverses the prefrontal area. A 30-second ramp-up period will be implemented at the commencement of the tDCS stimulation, followed by a 30-second ramp-down period at its conclusion.
  Interventions: Procedure: Exercise; Procedure: TDCS
- Exercise + ShamTDCS (Placebo Comparator): The device will be configured to produce an upward gradient for 30 seconds, identical to that used in the experimental group, followed by a downward gradient for another 30 seconds. Consequently, the control group will feel a similar tingling on their scalp as the experimental group. This stimulation will occur for a total of 60 seconds, which is insufficient to induce changes in cortical excitability. Studies have demonstrated that this approach effectively ensures patient blinding .
  Interventions: Procedure: Exercise; Procedure: ShamTDCS

INTERVENTIONS:
Procedure: Exercise — Structured treatment sessions, each lasting 30 minutes, will be organized into distinct blocks. In the initial phases, participants will engage in exercises emphasizing core stabilization and general strength training, with a particular focus on forced expiration as a technique to ensure the proper activation of the transversus abdominis muscle. This methodology aims to mitigate adverse effects associated with increased intra-abdominal pressure. To optimize the activation of the transversus abdominis, patients will be instructed to perform a forced expiration while concurrently drawing the navel inward and upward toward the spine, maintaining the lumbar spine in a neutral position. During the initial exercises, ultrasound imaging of the transversus abdominis will be employed as visual feedback, enabling patients to observe muscle thickening during forced expiration. This visual feedback enhances the accuracy of muscle activation and exercise technique. Exercises will be progressively s
Procedure: TDCS — The transcranial direct current stimulation (tDCS) protocol will involve the application of a continuous current for 30 minutes, with an intensity ranging from 1 to 1.5 mA, targeting the left dorsolateral prefrontal cortex (DLPFC) during each session. Two saline-soaked sponge electrodes, each measuring 35 cm², will be employed to ensure adequate skin contact. In accordance with the international 10-20 EEG electrode placement system, the anodal electrode will be positioned at the F3 location, specifically targeting the left DLPFC. The reference electrode will be placed above the left eye to facilitate efficient current flow through the prefrontal region of the brain. To enhance both safety and efficacy, a 30-second ramp-up and ramp-down period will be incorporated at the commencement and conclusion of the stimulation session. This methodology is intended to minimize potential adverse effects and ensure an optimal stimulation experience for participants.
  Arms: Exercise + TDCS
Procedure: ShamTDCS — The device will be configured to produce an upward gradient for 30 seconds, identical to that used in the experimental group, followed by a downward gradient for another 30 seconds. Consequently, the control group will feel a similar tingling on their scalp as the experimental group. This stimulation will occur for a total of 60 seconds, which is insufficient to induce changes in cortical excitability. Studies have demonstrated that this approach effectively ensures patient blinding.
  Arms: Exercise + ShamTDCS

SUMMARY:
Chronic spinal pain is a multifaceted condition frequently characterized by an absence of discernible structural causes, manifesting in symptoms such as significant disability and diminished quality of life. Persistent Spinal Pain Syndrome Type 2 (PSPS-T2) represents a common variant, implicating both peripheral and central nervous system mechanisms. This study investigates the synergistic effects of transcranial direct current stimulation (tDCS) in conjunction with motor control exercises on PSPS-T2 patients who have not responded to conventional treatments. A randomized controlled trial (RCT) will be conducted to compare an experimental group (tDCS + exercise) with a control group (exercise only), with the objective of enhancing functionality, alleviating pain levels, and improving psychological well-being. The findings may contribute to the development of more effective, patient-centered treatment strategies.

DETAILED DESCRIPTION:
Chronic spinal pain, characterized by persistent discomfort, frequently lacks discernible structural abnormalities and represents a complex, multifactorial condition. This disorder, manifested by symptoms such as lumbar pain, severe disability, diminished quality of life, and elevated unemployment rates, poses a substantial challenge for treatment. Therapeutic strategies encompass surgical intervention, pharmacological treatments, and conservative methods emphasizing exercise and behavioral therapies. However, the heterogeneous nature of these patients complicates both diagnosis and the assessment of clinical outcomes. Among the diagnostic terms for chronic spinal pain, Persistent Spinal Pain Syndrome (PSPS), particularly PSPS-T2, has garnered attention due to its high prevalence and recurrence in clinical pain management. The complexity of PSPS necessitates a multidisciplinary approach, with a recent shift towards patient-centered care, which has proven effective in reducing both direct and indirect costs associated with these patients. PSPS-T2 has the potential to affect a significant portion of the population, influenced by biological, psychological, and social components. The condition's neuroplasticity involves both peripheral and central mechanisms, which alter the central nervous system's state, contributing to the persistence of pain. Recent advancements in neuromodulatory strategies, such as non-invasive brain stimulation (NIBS), have shown promise in treating spinal pain, particularly in cases associated with neuropathic pain and comorbidities like depression. Additionally, motor control exercises and spinal stabilization have demonstrated efficacy in reducing pain and disability, supporting self-management and improving biopsychosocial beliefs. Combining exercise with NIBS may enhance outcomes, offering an alternative for patients resistant to conventional treatments. This study aims to evaluate the effects of combining neuromodulation (tDCS) with motor control exercises in PSPS-T2 patients. Specifically, we hypothesize that this combined intervention will lead to improvements in functionality, pain reduction, and psychological outcomes, benefiting patients who have not responded to other treatments. A randomized controlled trial (RCT) will be conducted with two groups: an experimental group receiving both tDCS and exercise, and a control group receiving only exercise. The primary objective is to assess baseline characteristics and the effects of the intervention on functionality, pain, psychosocial variables, depression, and quality of life. Secondary objectives include identifying clinical profiles and evaluating the impact of gender, age, and BMI on treatment outcomes. This study is expected to provide valuable insights into the efficacy of combined neuromodulation and exercise for managing PSPS-T2, with potential applications in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnostic of PSPS-T2
* Neuropathic pain (DNA4 ≥ 4)
* Patients older than 18 years
* ≥ 6 months with pain
* VAS score ≥ 7

Exclusion Criteria:

* Previous or programmed surgeries in abdominal area
* Pregnant or lactating
* Severe fractures or pathologies
* Spine structural deformity
* Neurologic or psychiatric issues

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
The Oswestry Disability Index (ODI) | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The Oswestry Disability Index (ODI) is the most widely used and validated assessment tool for low back pain. It is a self-administered questionnaire divided into ten sections designed to evaluate limitations in activities of daily living. Each section is scored on a scale from 0 to 5, with 5 indicating the highest level of disability. The total index score is calculated by dividing the sum of the section scores by the maximum possible score and multiplying by 100, yielding a percentage. The ODI has been validated in Spanish, demonstrating high sensitivity and specificity for functional assessment.

SECONDARY OUTCOMES:
Tampa Scale 11 (TSK-11) | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Kinesiophobia is defined as an excessive, irrational, and debilitating fear of physical movement and activity, stemming from a perceived vulnerability to a painful injury or reinjury. Fear of movement has been associated with disability in individuals with chronic pain. The Tampa Scale for Kinesiophobia (TSK) has been shown to predict the degree of disability in patients with chronic pain, with its scores correlating with depression, pain-related fear, and perceived pain intensity. Recently, the use of the TSK-11, a shortened version designed to identify fear-avoidance beliefs in musculoskeletal pain populations, has been recommended. The TSK-11 is scored between 11 and 44 points, with higher scores indicating greater fear of reinjury due to movement. The scale has demonstrated a 90% confidence interval and a reliability coefficient of 0.84.
Catastrophizing | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  Catastrophizing is understood as a set of negative emotional and cognitive processes that, by themselves, lead to an increase in pain symptoms and fatigue. It also involves a perceived helplessness in coping with pain and an inability to disengage from pain-related thoughts, whether in anticipation or recollection of the painful experience. Catastrophizing comprises three components: rumination, which refers to persistent worry and the inability to suppress thoughts related to pain; magnification, the tendency to exaggerate the unpleasantness of pain and amplify negative thoughts about pain relief; and helplessness, which arises from the perceived inability to cope with painful situations.
  To measure the level of catastrophizing in the present study, the Spanish validated version of the Pain Catastrophizing Scale (PCS) was used. This version demonstrates an internal consistency of 0.79 and a test-retest reliability of 0.84. The PCS is a self-administered questionnaire consisting of 1
SF-12 | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The SF-12 measures Health-Related Quality of Life (HRQoL) and comprises several dimensions: (a) physical functioning, (b) physical role, (c) emotional role, (d) social functioning, (e) bodily pain, and (f) vitality. Additionally, it includes two overarching dimensions that encompass the previous ones: (a) general health and (b) mental health. It is a widely used instrument in the healthcare field and has demonstrated satisfactory psychometric properties, including internal consistency and test-retest reliability.
Visual Analogue Scale (VAS) | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The VAS is considered the most representative scale and is regarded as the best option due to its simplicity and ease of use. The version employed in this study ranges from 0 to 10. This scale provides an effective tool for subjectively and discriminatively quantifying pain intensity. A score of 0 indicates no pain as reported by the individual, while 10 represents the worst imaginable pain. Due to these characteristics, the VAS has shown greater utility compared to descriptive or fixed-value scales. The VAS has demonstrated high reliability (Cronbach's α = 0.97) [95% CI = 0.96 to 0.98].
DN4 Questionnaire | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The DN4 is one of the most sensitive questionnaires for diagnosing neuropathic pain, demonstrating a high capacity to distinguish between neuropathic and nociceptive pain. The DN4 has been validated in patients with low back pain (LBP) due to disc herniation, spinal stenosis, degenerative disc disease, spinal pain, lumbar spine degeneration, spinal surgery, and lumbar scoliosis. A DN4 cutoff score of 4 yielded a sensitivity of 80% and a specificity of 92% for the diagnosis of neuropathic pain in individuals with LBP. Each patient was asked to describe their pain using the first seven descriptors of neuropathic pain in the DN4, in order to calculate the DN4 interview subscore (range: 0-7).
Beck Depression Inventory | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  The Beck Depression Inventory - Second Edition (BDI-II) is a self-report instrument consisting of 21 items used to measure the severity of depression in adults and adolescents over the age of 13. This version of the inventory (BDI-II) was developed to assess symptoms corresponding to the criteria for diagnosing depressive disorders outlined in the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV; 1994)
The Chronic Pain Self-Efficacy Questionnaire by Martín-Aragón | Pre-treatment, 1-month follow-up, 3-month follow-up, 6-month follow-up
  For this reason, a scale was designed to evaluate self-efficacy expectations regarding symptom management, physical functioning, and pain control. The Chronic Pain Self-Efficacy Questionnaire by Martín-Aragón et al. (1998), validated in Spanish, was used, as its validation results are comparable to those of the original scale by Anderson et al. (1995). This version demonstrates high internal consistency (α = 0.87). The questionnaire consists of 19 items, uses a Likert-type scale, and has a response range from 0 to 10, where 0 represents feeling completely incapable, 5 moderately capable, and 10 fully capable.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic Univerity of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sebaaly A, Lahoud MJ, Rizkallah M, Kreichati G, Kharrat K. Etiology, Evaluation, and Treatment of Failed Back Surgery Syndrome. Asian Spine J. 2018 Jun;12(3):574-585. doi: 10.4184/asj.2018.12.3.574. Epub 2018 Jun 4. PMID 29879788
- [Background] Bursali C, Ozkan FU, Kaysin MY, Dortcan N, Aktas I, Kulcu DG. Effectiveness of Repetitive Transcranial Magnetic Stimulation in Patients With Failed Back Surgery Syndrome: A Double-Blind Randomized Placebo-Controlled Study. Pain Physician. 2021 Jan;24(1):E23-E30. PMID 33400434
- [Derived] Huertas-Ramirez B, Jaenada-Carrilero E, Belda-Antoli M, Leal-Garcia J, Alonso-Martin M, Mahiques-Sanchis A, Benlloch-Garcia A, Falaguera-Vera F, Vicente-Mampel J. Patient-Centered Chronic Spinal Pain Management Using Exercise and Neuromodulation: Study Protocol for a Randomized Controlled Trial. Healthcare (Basel). 2025 Nov 24;13(23):3032. doi: 10.3390/healthcare13233032. PMID 41373250